CLINICAL TRIAL: NCT02837601
Title: A Single Center, Prospective, Randomized, Controlled Study To Evaluate Physician Preference Related To The Use Of The Surgiquest Airseal® Insufflation System (AIS) At Low Vs. Higher Pressure For The Management Of Pneumoperitoneum
Brief Title: Pneumoperitoneum Management With SurgiQuest AirSeal® at Low vs. Higher Pressure
Acronym: PRESSURE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Principal Investigator, Todd Ponsky, MD, Akron Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRESSURE
Record Dates: First submitted 2015-01-13; First posted 2016-07-19 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Shoulder Pain
Keywords: Laparoscopic surgical procedures; Shoulder Pain; Abdominal Pain; Pediatrics
MeSH Terms: conditions — Shoulder Pain; Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- LOW AIS Pressure AirSeal® (Other): AIS with an insufflation pressure target of 9mmHg ±1mmHg
  Interventions: Device: AirSeal® Insufflation System (AIS)
- HIGH AIS Pressure AirSeal® (Other): AIS with an insufflation pressure target of 15mmHg ±1mm
  Interventions: Device: AirSeal® Insufflation System (AIS)

INTERVENTIONS:
Device: AirSeal® Insufflation System (AIS) — The AirSeal® System consists of an insufflation, filtration, and recirculation system (AirSeal® iFS), a triple lumen filtered tube set, and a valve free trocar (AirSeal® Access Port). The device enables peritoneal access with a novel mechanism to maintain pneumoperitoneum without a mechanical seal. Specifically, the AirSeal® System creates a pressure barrier within the proximal housing of the cannula which acts as an invisible seal to maintain pneumoperitoneum during the course of surgery. It utilizes a re-circulation and filtration control unit (AirSeal® iFS) designed specifically for the AirSeal® Access Port to create and maintain the pressure barrier.

SUMMARY:
A prospective, randomized, controlled single-center clinical Study designed to evaluate Physician Preference related to the use of the SurgiQuest AirSeal® Insufflation System (AIS) at low vs. higher pressures for the Management of pneumoperitoneum. Subjects will be randomized in a 1:1 treatment device to control ratio into one of two (2) different study arms:

1. AIS with an insufflation pressure target of 9mmHg ±1mmHg; or
2. AIS with an insufflation pressure target of 15mmHg ±1mmHg.

DETAILED DESCRIPTION:
The study is designed and powered to demonstrate superiority of the AIS at low pressure vs. at higher pressure on a single key effectiveness measure: Incidence of shoulder pain. Patients will be randomized 1:1 to either AIS with an insufflation pressure target of 9mmHg ±1mmHg or to AIS with an insufflation target pressure of 15mmHg ±1mmHg.

Secondary outcome measures include severity of shoulder pain measured using a VAS scale and medication use, length of hospital stay, aspects of anesthesia management including end tidal CO2 and the frequency of adverse events. These outcomes will be evaluated in a controlled population undergoing laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric subjects (<21 years of age)
2. > 20 kg in weight;
3. Capable and willing to provide parental Informed Consent and patient Assent;
4. Acceptable candidate for laparoscopic surgery;

Exclusion Criteria:

1. Active cutaneous infection or inflammation;
2. Pre-existing immunodeficiency disorder and/or chronic use of systemic steroids;
3. Uncontrolled diabetes mellitus
4. Known, significant history of bleeding diathesis, coagulopathy, von Willebrand's disease or current platelet count < 100,000 cells/mm3, baseline INR(international normalized ratio) ≥1.8, or fibrinogen level less than 150 mg/dl (if received a fibrinolytic agent within prior 24 hours);
5. Severe co-existing morbidities having a life expectancy of less than 30 days;
6. Currently involved in any other investigational clinical Studies;
7. Significant anemia with a hemoglobin level less than 10 g/dL or a hematocrit less than 30%;
8. Females who are pregnant, planning to become pregnant within 3 months of the procedure, or lactating;
9. Extreme morbid obesity (BMI greater than 45 kg/m2)
10. Patients presenting with Ascites

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Post-operative shoulder pain | Post-operative shoulder pain will be assessed at 24 hours after surgery, or at the time of discharge, whichever comes first.
  Severity of shoulder pain, which will be measured using the Face, Legs, Activity, Cry, Consolability (FLACC) scale or Wong-Baker FACES Pain Rating Scale, whichever is deemed more appropriate by the clinician assessing the patient.

SECONDARY OUTCOMES:
Pain severity and trend | Pain will be assessed at least daily from the immediate post-operative period until discharge from the hospital, up to 10 days.
  Severity of shoulder pain, back pain, abdominal pain. Pain will be measured using the Face, Legs, Activity, Cry, Consolability (FLACC) scale or Wong-Baker FACES Pain Rating Scale, whichever is deemed more appropriate by the clinician assessing the patient.
Pressure stability | During procedure
  Stability of intra-abdominal pressure
Ease of anesthesia management | During procedure
  Excessively high peak and/or mean airway pressures. Anesthesiologist reported difficulty with ventilation.
Length of recovery room stay | Post-anesthesia care unit (PACU) discharge, up to 24 hours.
  A measure of time the patient spends in the post-anesthesia recovery area
Length of Stay (LOS) | Until the time of hospital discharge, up to 10 days.
  The length of hospital stay associated with the surgery. This will be assessed through study completion. It is anticipated to be less than 10 days but could potentially exceed this length as the length of stay cannot always be predicted and there is no upper limit on hospital length of stay.
Procedural related Adverse Events/ Serious Adverse Events (AEs/ SAEs? | During hospital stay up to 30 days
Rate of device-related events | During procedure

CONTACTS AND LOCATIONS:
Overall Officials: Todd Ponsky, MD, Principal Investigator — Akron Children's Hospital
Locations (1):
- Children's Hospital Medical Center of Akron, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurusamy KS, Samraj K, Davidson BR. Low pressure versus standard pressure pneumoperitoneum in laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD006930. doi: 10.1002/14651858.CD006930.pub2. PMID 19370662
- [Background] Hua J, Gong J, Yao L, Zhou B, Song Z. Low-pressure versus standard-pressure pneumoperitoneum for laparoscopic cholecystectomy: a systematic review and meta-analysis. Am J Surg. 2014 Jul;208(1):143-50. doi: 10.1016/j.amjsurg.2013.09.027. Epub 2014 Jan 16. PMID 24503370